CLINICAL TRIAL: NCT02060799
Title: European Dyspnoea Survey in the EMergency Departments
Acronym: EuroDEM
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Said LARIBI, MD, PhD., Principal Investigator, Hopital Lariboisière
Other Study IDs: HLariboisiere
Record Dates: First submitted 2014-02-09; First posted 2014-02-12 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Dyspnea; Emergencies
Keywords: Dyspnea; Emergency Service, Hospital; prognosis; Fatal Outcome; Epidemiology
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Braunwald defines dyspnoea as an abnormally uncomfortable awareness of breathing. Breathing discomfort, and its varying degrees of severity, is the one of the most disturbing symptoms patients can experience; and it is one of the main complaints in the patients presenting to the Emergency Department (ED). Dyspnea has a variety of underlying etiologies, like cardiac, pulmonary or metabolic etiologies or a combination of them, since several diseases can cause dyspnea like for instance heart failure (HF), asthma and chronic obstructive pulmonary disease (COPD).

Acute heart failure syndrome (AHFS) is collectively defined as a gradual or rapid change in heart failure (HF) signs and symptoms resulting in a need for urgent therapy. Heart failure (HF) is one of the most important causes of morbidity and mortality in the industrialized world. The prevalence of symptomatic HF is estimated to range from 0.4 to 2.0% in general European population. The incidence increases rapidly with age, and in Europe. Characteristics, clinical presentation, treatment, and outcomes of HF patients admitted to hospital have been adequately described, in Europe and in the United States. The Euro Heart Failure Survey (EHFS) I with 11 327 patients described the demographics of acutely hospitalized HF patients. The ADHERE registry has data on over 100 000 hospitalizations for AHF from the USA. In-hospital mortality was 4 and 7%, in ADHERE and EHFS I, respectively.

This same sensation of breathlessness is what also drives patients with asthma and chronic obstructive pulmonary disease (COPD) to the ED. Chronic obstructive pulmonary disease (COPD) exacerbation accounts for approximately 1.5 million ED visits in the United States per year. It is the third most common cause of hospitalization, with an estimated 726 000 hospitalizations in 2000 in the USA. Previous studies have demonstrated important differences between guideline recommendations and actual management of COPD exacerbation, either in the ED or during hospitalization.

The diagnosis in front of a dyspneic patient in the ED remains a challenge, because of a low sensitivity of the clinical signs associated with the aging of the population and the variety of underlying diseases. Little is known about the Epidemiology of dyspneic patients in the ED at the European level. Diagnosis, prevalence and treatment of the patients may vary among European countries.

DETAILED DESCRIPTION:
MAIN OBJECTIVES

* Epidemiologic description of patients presenting to the ED with shortness of breath as main complaint.
* Description of current management in the ED of patients presenting to the ED with shortness of breath as main complaint.

SECONDARY OBJECTIVES

* Sub analysis of ED discharged patients versus admitted patients for characteristics, comparison to recommended care and re-ED visit.
* Determine clinical and/or biological criteria to distinguish between:

  * Patients who are treated as outpatients and admitted patients.
  * Patients hospitalized in ward and patients admitted to intensive care units (CCU and ICU)
* Prognostic prediction, using clinical and biochemical data
* To determine if ED patients treated for acute heart failure differ from those admitted to hospital.
* Comparison of European data characteristics, investigation, treatment and outcome to similar data in other part of the world.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting to the Emergency Department with Dyspnea as main complaint
* 18 years or older

Exclusion Criteria:

* No acceptance to participate from the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to the Emergency Department with Dyspnea as main complaint during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2156 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  All cause mortality will be evaluated 30 days after ED visit.

SECONDARY OUTCOMES:
All cause rehospitalization | 30 days

OTHER OUTCOMES:
ED visit | 30 days
  New ED visit during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Said LARIBI, MD, PhD, Principal Investigator — Lariboisière Hospital, EuSEM
Locations (10):
- Country: Belgium, Brussels, Belgium
- Country: Finland, Helsinki, Finland
- Country: France, Paris, France
- Country: Germany, Nuremberg, Germany
- Country: Italy, Rome, Italy
- Country: Netherlands, Amsterdam, Netherlands
- Country: Romania, Cluj-Napoca, Romania
- Country: Spain, Santander, Spain
- Country: Turkey, Ankara, Turkey (Türkiye)
- Country: United Kingdom, Manchester, United Kingdom